CLINICAL TRIAL: NCT00905450
Title: Evaluation of BOL-303242-X Versus Vehicle for the Treatment of Inflammation Following Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 588
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Cataract; Inflammation
Keywords: Surgery
MeSH Terms: conditions — Cataract; Inflammation | interventions — R-1,1,1-trifluoro-4-(5-fluoro-2,3-dihydrobenzofuran-7-yl)-4-methyl-2-(((2-methyl-5-quinolyl)amino)methyl)pentan-2-ol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOL-303242-X (Experimental): BOL-303242-X (Mapracorat)
  Interventions: Drug: BOL-303242-X
- Vehicle (Placebo Comparator): Vehicle for BOL-303242-X (Mapracorat)
  Interventions: Drug: Vehicle for BOL-303242-X

INTERVENTIONS:
Drug: BOL-303242-X — Medication instilled into the study eye, subjects randomized to various drug concentrations and dose schedules.
  Other Names: Mapracorat
  Arms: BOL-303242-X
Drug: Vehicle for BOL-303242-X — Medication instilled into the study eye, subjects randomized to various drug dose schedules.
  Arms: Vehicle

SUMMARY:
This clinical study is being conducted to identify the most effective drug concentration and dose frequency of BOL-303242-X (Mapracorat) ophthalmic suspension, for the treatment of inflammation following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age on the date the Informed Consent Form (ICF) is signed and with the capacity to voluntarily provide consent.
* Subjects must be able to understand and provide written consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide authorization as appropriate for local privacy regulations.
* Subjects who are candidates for cataract surgery.
* Subjects who are not of childbearing potential or female subjects who have a negative urine pregnancy test result at screening.
* Subjects must be able and willing to comply with all treatment and follow- up procedures.

Exclusion Criteria:

* Subjects who have known hypersensitivity or contraindication to the study drug(s) or their components.
* Subjects who have a history or presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result of the study.
* Subjects who have a severe/serious ocular condition, or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% Twice a Day: BOL-303242-X ophthalmic suspension 1% Twice a Day
- 2% Once a Day: BOL-303242-X ophthalmic suspension 2% Once a Day
- 2% Twice a Day: BOL-303242-X ophthalmic suspension 2% Twice a Day
- 2% Four Times a Day: BOL-303242-X ophthalmic suspension 2% Four times a Day
- 3% Once a Day: BOL-303242-X ophthalmic suspension 3% Once a Day
- 3% Twice a Day: BOL-303242-X ophthalmic suspension 3% Twice a Day
- 3% Four Times a Day: BOL-303242-X ophthalmic suspension 3% Four times a Day
- Vehicle: Vehicle for BOL-303242-X ophthalmic suspension
Period: Overall Study
Arm/Group | 1% Twice a Day | 2% Once a Day | 2% Twice a Day | 2% Four Times a Day | 3% Once a Day | 3% Twice a Day | 3% Four Times a Day | Vehicle
Started | 60 | 28 | 28 | 60 | 59 | 60 | 60 | 60
Completed | 59 | 27 | 28 | 60 | 59 | 58 | 58 | 59
Not Completed | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Twice a Day | 2% Once a Day | 2% Twice a Day | 2% Four Times a Day | 3% Once a Day | 3% Twice a Day | 3% Four Times a Day | Vehicle | Total
Number analyzed (Participants) | 60 | 28 | 28 | 60 | 59 | 60 | 60 | 60 | 415
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (12.0) | 67.9 (10.9) | 68.9 (10.5) | 69.5 (7.1) | 68.2 (10.8) | 67.3 (10.7) | 68.5 (10.3) | 67.1 (10.8) | 67.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 15 | 15 | 34 | 30 | 32 | 31 | 32 | 222
  Male | 27 | 13 | 13 | 26 | 29 | 28 | 29 | 28 | 193

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells.
Description: Anterior chamber (AC) cells will be assessed using a 0 to 4 grading scale by an ophthalmologist using slip lamp biomicroscopy. A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens was performed without pupil dilation. Accumulation of white blood cells in aqueous was assessed. Pigment cells and red blood cells are to be ignored. The grades were defined as: 0 = No cells seen; 1 = 1 - 5 cells; 2 = 6 - 15 cells; 3 = 16 - 30 cells; 4 = >30 cells. Complete resolution of AC cells was defined as Grade 0.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Twice a Day | 2% Once a Day | 2% Twice a Day | 2% Four Times a Day | 3% Once a Day | 3% Twice a Day | 3% Four Times a Day | Vehicle
Number analyzed (Participants) | 60 | 28 | 28 | 60 | 59 | 60 | 60 | 60
Participants | 35 | 19 | 15 | 47 | 42 | 45 | 42 | 30

2. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Flare.
Description: A slit lamp examination of the lids, conjunctiva, limbus, cornea, anterior chamber, vitreous, and lens will be performed without pupil dilation. Scattering of a slit lamp light beam when directed into the anterior chamber (Tyndall effect). The grades for flare were 0=None to 4=Very Severe effect. Complete resolution of AC flare was defined as Grade 0.
Time Frame: 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1% Twice a Day | 2% Once a Day | 2% Twice a Day | 2% Four Times a Day | 3% Once a Day | 3% Twice a Day | 3% Four Times a Day | Vehicle
Number analyzed (Participants) | 60 | 28 | 28 | 60 | 59 | 60 | 60 | 60
Participants | 15 | 6 | 7 | 18 | 21 | 23 | 18 | 11

ADVERSE EVENTS:
Time Frame: 18 days
Arm/Group | 1% Twice a Day | 2% Once a Day | 2% Twice a Day | 2% Four Times a Day | 3% Once a Day | 3% Twice a Day | 3% Four Times a Day | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/28 | 0/28 | 0/60 | 1/59 | 1/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 43/60 | 20/28 | 7/28 | 18/60 | 11/59 | 25/60 | 21/60 | 37/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Twice a Day (N=60) | 2% Once a Day (N=28) | 2% Twice a Day (N=28) | 2% Four Times a Day (N=60) | 3% Once a Day (N=59) | 3% Twice a Day (N=60) | 3% Four Times a Day (N=60) | Vehicle (N=60)
Cystoid macular edema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subretinal neovascularization (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Twice a Day (N=60) | 2% Once a Day (N=28) | 2% Twice a Day (N=28) | 2% Four Times a Day (N=60) | 3% Once a Day (N=59) | 3% Twice a Day (N=60) | 3% Four Times a Day (N=60) | Vehicle (N=60)
Headache (Nervous system disorders) | 2 | 0 | 0 | 4 | 1 | 1 | 0 | 0
Eye pain (Eye disorders) | 7 | 4 | 2 | 0 | 3 | 2 | 2 | 6
Photophobia (Eye disorders) | 7 | 4 | 0 | 1 | 1 | 4 | 4 | 5
AC Inflammation (Eye disorders) | 2 | 1 | 0 | 2 | 1 | 3 | 2 | 4
Ocular hyperaemia (Eye disorders) | 5 | 1 | 0 | 1 | 1 | 2 | 3 | 2
Lacrimation increased (Eye disorders) | 3 | 2 | 0 | 2 | 1 | 2 | 2 | 2
Corneal edema (Eye disorders) | 2 | 4 | 1 | 1 | 0 | 1 | 1 | 3
Foreign body sensation in eyes (Eye disorders) | 4 | 0 | 0 | 1 | 0 | 2 | 3 | 2
Dry eye (Eye disorders) | 3 | 2 | 0 | 1 | 0 | 2 | 1 | 0
Eye pruritis (Eye disorders) | 4 | 2 | 0 | 0 | 1 | 1 | 1 | 0
Iritis (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4
Conjunctival hyperemia (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
AC Flare (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Ciliary hyperemia (Eye disorders) | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 0
Intraocular pressure increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.